CLINICAL TRIAL: NCT06943885
Title: Comparison of 5G Mobile Stroke Unit to Standard Management by Emergency Medical Services For Acute Ischemic Stroke Treatment：A Multicenter, Prospective, Open-label, Blinded Endpoint , Week-wise Randomized, Controlled Trial
Brief Title: Comparison of 5G-Mobile Stroke Unit With Standard EMS for Acute Ischemic Stroke
Acronym: 5G-MSU-FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Emergency Medical Center (Other)
Responsible Party: Principal Investigator, Dou Li, Principal Investigator, Beijing Emergency Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023ZD0503802
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5G Mobile Stroke Unit Management (Experimental): AIS patients treated in the Mobile Stroke Unit
  Interventions: Other: 5G Mobile Stroke Unit Management
- Standard Management (Active Comparator): AIS patients receiving standard management
  Interventions: Other: Standard Management

INTERVENTIONS:
Other: 5G Mobile Stroke Unit Management — 5G MSU is a specialized stroke ambulance equipped with point of care lab, CT scanner, Telemedicine, allowing patients to receive intravenous thrombolysis.
  Arms: 5G Mobile Stroke Unit Management
Other: Standard Management — A regular ambulance. The standard management by EMS includes Electrocardiographic（ECG）monitoring, blood glucose management, airway, respiration, and blood pressure control, complication management, intravenous access establishment and other emergency measures.
  Arms: Standard Management

SUMMARY:
While Mobile Stroke Units (MSUs) are considered as a relatively new model for acute stroke treatment, 5G Mobile Stroke Units (5G MSUs) have already come into service for stroke treatment in some parts of China. Since limited evidence has been found to suggest their advantages over conventional Emergency Medical Services (EMS), well-conducted clinical studies are required to further assess their effectiveness and safety. This study aims to evaluate whether 5G MSUs outperform standard management (SM) by EMS in terms of functional outcomes of acute ischemic stroke (AIS) patients within 4.5 hours after symptom onset in urban and rural areas of China.

DETAILED DESCRIPTION:
This Multicenter, Prospective, Open-label, Blinded Endpoint , Week-wise Randomized, Controlled trial will allocate patients to one of two study arms for the analyses：one group will receive pre-hospital diagnosis and treatment in a 5G MSU followed by transfer to a Comprehensive Stroke Center (CSC) Emergency Department (ED) for further management; the other group will undergo standard pre-hospital triage with subsequent transport by EMS to a CSC ED for evaluation and treatment. The main criteria to enroll a patient into the study include: a. history and physical/neurological examination consistent with acute stroke, b. age≥18, c. last seen normal within 4hr 30 min of symptom onset, d. pre-stroke modified Rankin scale ≤3 (Being able to ambulate), e. no Recombinant tissue Plasminogen Activator（rt-PA）or Tenecteplase（TNK）exclusions per guidelines, prior to CT scan or baseline labs and f. informed consent obtained from patient (if competent) or legal representative. The primary outcome was the distribution of modified Rankin Scale (mRS) scores (a disability score ranging from 0, no neurological deficits, to 6, death) at 3 months.

It is hypothesized that the 5G MSU pathway, compared to EMS, can enable earlier evaluation and treatment of AIS patients within 4.5 hours of onset, thereby improving functional outcomes three months after stroke while ensuring safety. The successful completion of this project will provide data on important outcomes and costs associated with the use of 5G MSU vs SM in China that will help determine the value of integrating 5G MSUs into the pre-hospital environment in this country.

ELIGIBILITY:
Inclusion Criteria:

1. History and physical/neurological examination consistent with acute stroke.
2. Age≥18.
3. Last seen normal within 4hr 30 min of symptom onset.
4. Pre-stroke modified Rankin scale ≤3（Being able to ambulate）.
5. No rt-PA/TNK exclusions per guidelines, prior to CT scan or baseline labs.
6. Informed consent obtained from patient (if competent) or legal representative.

Exclusion Criteria:

1. Malignant or other severe primary disease with life expectancy <1 year.
2. Participation in other interventional randomized clinical trials within 3 months before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 90 days (±7 days) from date of enrollment
  Assessment of functional outcome using the Modified Rankin Scale (mRS), a disability scale that ranges from 0 (no symptoms) to 6 (death), with higher scores indicating worse functional outcomes.

SECONDARY OUTCOMES:
Proportion of patients achieving mRS 0-1 | 90 days (±7 days) from date of enrollment
  Excellent functional outcome (Modified Rankin Scale score, mRS 0-1)
Intravenous Thrombolysis rate（A） | up to 4.5 hours from symptom onset
  Proportion of participants ultimately treated with Intravenous Thrombolysis（IVT）within 4.5 hours
Intravenous Thrombolysis rate（B） | up to 1 hours from symptom onset
  Proportion of participants ultimately treated with IVT within 60 minutes.
Endovascular treatment rate | up to 24 hours from symptom onset
  Proportion of participants ultimately treated with Endovascular treatment（EVT）
Diagnosis and treatment times (A) | up to 4.5 hours from symptom onset
  Onset-to-IVT time
Diagnosis and treatment times (B) | up to 4.5 hours from symptom onset
  Onset-to-IVT decision time
Diagnosis and treatment times (C) | up to 24 hours from symptom onset
  Onset-to-EVT time
Diagnosis and treatment times (D) | up to 4.5 hours from symptom onset
  Alarm-to-IVT time
Diagnosis and treatment times (E) | up to 4.5 hours from symptom onset
  Alarm-to-IVT decision time
Diagnosis and treatment times (F) | up to 24 hours from symptom onset
  Alarm-to-EVT time
Diagnosis and treatment times (G) | up to 24 hours from symptom onset
  Emergency Department（ED）arrival-to-EVT time
Quality of life（A） | 90 days (±7 days) from date of enrollment
  Assessment with European Quality of Life - 5 Dimensions (EQ-5D)
Quality of life（B） | 90 days (±7 days) from date of enrollment
  Assessment with Barthel Index
Cost-Effectiveness(A) | 12 month (±14 days) from date of enrollment
  Cost-Effectiveness as measured by patient Quality-Adjusted Life Year（QALYs）
Cost-Effectiveness (B) | up to hospital discharge
  Cost-Effectiveness as measured by post-stroke healthcare utilization
Rate of symptomatic intracranial hemorrhage（ECASS III） | 36 hours from time of enrollment
  The incidence of symptomatic intracranial hemorrhage (sICH) , According to the European Cooperative Acute Stroke Study III
In-hospital mortality rate | 7 days (±1 day) /discharge from date of enrollment
  Frequency of patients dying within the duration of the hospital stay after admission for stroke
All-cause mortality rate | 90 days (±7 days) from date of enrollment
  All-cause mortality rate at 90±7 days
Rate of stroke mimics and transient ischemic attacks | up to hospital discharge
  The incidence of stroke mimics and transient ischemic attacks (TIAs)

CONTACTS AND LOCATIONS:
Overall Officials: Dou Li, MD, Principal Investigator — Beijing Emergency Medical Center
Locations (1):
- Beijing Emergency Medical Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No